CLINICAL TRIAL: NCT03021499
Title: A Randomized, Controlled Double-blind Study Comparing the Efficacy and Safety of Voclosporin (23.7 mg Twice Daily) With Placebo in Achieving Renal Response in Subjects With Active Lupus Nephritis
Brief Title: Aurinia Renal Response in Active Lupus With Voclosporin
Acronym: AURORA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aurinia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUR-VCS-2016-01
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Results first posted 2021-06-16 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Lupus Nephritis
Keywords: lupus nephritis; calcineurin inhibitors; voclosporin
MeSH Terms: conditions — Lupus Nephritis | interventions — voclosporin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Voclosporin (Experimental): oral, 23.7 mg twice daily (BID)
  Interventions: Drug: Voclosporin
- Placebo Oral Capsule (Placebo Comparator): Voclosporin placebo, oral, 3 capsules twice daily (BID)
  Interventions: Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Voclosporin — calcineurin inhibitor
  Other Names: ISA247
  Arms: Voclosporin
Drug: Placebo Oral Capsule — matching placebo capsule
  Arms: Placebo Oral Capsule

SUMMARY:
The purpose of this study is to assess the efficacy of voclosporin compared with placebo in achieving renal response after 52 weeks of therapy in subjects with active lupus nephritis.

DETAILED DESCRIPTION:
The aim of the current study is to investigate whether voclosporin, added to the standard of care treatment in active lupus nephritis (LN), is able to reduce disease activity over a treatment period of 52 weeks. The background therapy will be mycophenolate mofetil (MMF) and initial treatment with IV methylprednisolone, followed by a reducing course of oral corticosteroids. Subjects with active, flaring LN will be eligible to enter the study. They are required to have a diagnosis of LN according to established diagnostic criteria and clinical and biopsy features suggestive of active nephritis. Efficacy will be assessed by the ability of the drug combination to reduce the level of proteinuria (as measured by Urine Protein Creatinine Ratio (UPCR)) while demonstrating an acceptable safety profile.

ELIGIBILITY:
Key Inclusion Criteria:

- Subjects with evidence of active nephritis, defined as follows:

* Kidney biopsy result within 2 years prior to screening indicating Class III, IV-S, IV-G (alone or in combination with Class V), or Class V LN with a doubling or greater increase of UPCR within the last 6 months to a minimum of ≥1.5 mg/mg for Class III/IV or to a minimum of ≥2 mg/mg for Class V at screening. Biopsy results over 6 months prior to screening must be reviewed with a medical monitor to confirm eligibility.

OR

* Kidney biopsy result within 6 months prior to screening indicating Class III, IV-S or IV-G (alone or in combination with Class V) LN with a UPCR of ≥1.5 mg/mg at screening.

OR

* Kidney biopsy result within 6 months prior to screening indicating Class V LN and a UPCR of ≥2 mg/mg at screening.

  * Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test at baseline.

Exclusion Criteria:

* Estimated glomerular filtration rate (eGFR) of ≤45 mL/minute at screening.
* Current or medical history of:

  * Congenital or acquired immunodeficiency.
  * In the opinion of the Investigator, clinically significant drug or alcohol abuse within 2 years prior to screening.
  * Malignancy within 5 years of screening, with the exception of basal and squamous cell carcinomas treated by complete excision.
  * Lymphoproliferative disease or previous total lymphoid irradiation.
  * Severe viral infection or known HIV infection.
  * Active tuberculosis (TB), or known history of TB/evidence of old TB if not taking prophylaxis with isoniazid.
* Other known clinically significant active medical conditions, such as:

  * Severe cardiovascular disease, liver dysfunction or chronic obstructive pulmonary disease or asthma requiring oral steroids or any other overlapping autoimmune condition for which the condition or the treatment of the condition may affect the study assessments or outcomes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2019-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir Parikh, MD, Principal Investigator — Ohio State University
Locations (172):
- United States (50):
  - AURORA Investigative Center, Huntsville, Alabama
  - AURORA Investigative Center, Phoenix, Arizona
  - AURORA Investigative Center, Beverly Hills, California
  - AURORA Investigative Center, Los Angeles, California
  - AURORA Investigative Center, Palo Alto, California
  - AURORA Investigative Center, Thousand Oaks, California
  - AURORA Investigative Center, Torrance, California
  - AURORA Investigative Center, Aurora, Colorado
  - AURORA Investigative Center, Denver, Colorado
  - AURORA Investigative Center, New Haven, Connecticut
  - AURORA Investigative Center, Clearwater, Florida
  - AURORA Investigative Center, DeBary, Florida
  - AURORA Investigative Center, Fort Lauderdale, Florida
  - AURORA Investigative Center, Fort Myers, Florida
  - AURORA Investigative Center, Miami, Florida
  - AURORA Investigative Center, Orlando, Florida
  - AURORA Investigative Center, Winter Park, Florida
  - AURORA Investigative Center, Atlanta, Georgia
  - AURORA Investigative Center, Columbus, Georgia
  - AURORA Investigative Center, Lawrenceville, Georgia
  - AURORA Investigative Center, Chicago, Illinois
  - AURORA Investigative Center, Louisville, Kentucky
  - AURORA Investigative Center, Baton Rouge, Louisiana
  - AURORA Investigative Center, New Orleans, Louisiana
  - AURORA Investigative Center, Boston, Massachusetts
  - AURORA Investigative Center, Detroit, Michigan
  - AURORA Investigative Center, Grand Blanc, Michigan
  - AURORA Investigative Center, Rochester, Minnesota
  - AURORA Investigative Center, St Louis, Missouri
  - AURORA Investigative Center, Las Vegas, Nevada
  - AURORA Investigative Center, Newark, New Jersey
  - AURORA Investigative Center, Great Neck, New York
  - AURORA Investigative Center, New York, New York
  - AURORA Investigative Center, Syracuse, New York
  - AURORA Investigative Center, Chapel Hill, North Carolina
  - AURORA Investigative Center, Charlotte, North Carolina
  - AURORA Investigative Center, Greenville, North Carolina
  - AURORA Investigative Center, New Bern, North Carolina
  - AURORA Investigative Center, Cleveland, Ohio
  - AURORA Investigative Center, Columbus, Ohio
  - AURORA Investigative Center, Oklahoma City, Oklahoma
  - AURORA Investigative Center, Charleston, South Carolina
  - AURORA Investigative Center, Chattanooga, Tennessee
  - AURORA Investigative Center, Hendersonville, Tennessee
  - AURORA Investigative Center, Beaumont, Texas
  - AURORA Investigative Center, Dallas, Texas
  - AURORA Investigative Center, El Paso, Texas
  - AURORA Investigative Center, Houston, Texas
  - AURORA Investigative Center, Arlington, Virginia
  - AURORA, Richmond, Virginia
- Argentina (5):
  - AURORA Investigative Center, Buenos Aires
  - AURORA Investigative Center, Caba
  - AURORA Investigative Center, Córdoba
  - AURORA Investigative Center, La Plata
  - AURORA Investigative Center, San Miguel de Tucumán
- Belarus (3):
  - AURORA Investigative Cener, Minsk
  - AURORA Investigative Center, Minsk
  - AURORA Investigative Center, Vitebsk
- Brazil (4):
  - AURORA Investigative Center, Curitiba
  - AURORA Investigative Center, Porto Alegre
  - AURORA Investigative Center, Salvador
  - AURORA Investigative Center, São Paulo
- Bulgaria (5):
  - AURORA Investigative Center, Plovdiv
  - AURORA Investigative Center, Smolyan
  - AURORA Investigative Center, Sofia
  - AURORA Investigative Center, Stara Zagora
  - AURORA Investigative Center, Vidin
- Canada (3):
  - AURORA Investigative Center, Edmonton, Alberta
  - AURORA Investigative Center, Montreal, Quebec
  - AURORA Investigative Center, Toronto
- Chile (3):
  - AURORA Investigative Center, Santiago
  - AURORA Investigative Center, Temuco
  - AURORA Investigative Center, Valdivia
- Colombia (4):
  - AURORA Investigative Center, Barranquilla
  - AURORA Investigative Center, Bogotá
  - AURORA Investigative Center, Bucaramanga
  - AURORA Investigative Center, Zipaquirá
- AURORA Investigative Center, San José, Costa Rica
- Croatia (2):
  - AURORA Investigative Center, Osijek
  - AURORA Investigative Center, Zagreb
- Dominican Republic (2):
  - AURORA Investigative Center, Santiago de los Caballeros
  - AURORA Investigative Center, Santo Domingo
- AURORA Investigative Center, Guatemala City, Guatemala
- Japan (12):
  - AURORA Investigative Center, Kita, Osaka
  - AURORA Investigative Center, Chiba
  - AURORA Investigative Center, Hiroshima
  - AURORA Investigative Center, Ishikawa
  - AURORA Investigative Center, Kita-ku
  - AURORA Investigative Center, Kitakyushu
  - AURORA Investigative Center, Maebashi
  - AURORA Investigative Center, Nagasaki
  - AURORA Investigative Center, Niigata
  - AURORA Investigative Center, Sapporo
  - AURORA Investigative Center, Sendai
  - AURORA Investigative Center, Tokyo
- AURORA Investigative Center, Kuala Lumpur, Malaysia
- Mexico (10):
  - AURORA Investigative Center, Baja California
  - AURORA Investigative Center, Coahuila
  - AURORA Investigative Center, Guadalajara
  - AURORA Investigative Center, León
  - AURORA Investigative Center, Mexico City
  - AURORA Investigative Center, Mérida
  - AURORA Investigative Center, Monclova
  - AURORA Investigative Center, Oaxaca City
  - AURORA Investigative Center, San Luis Potosí City
  - AURORA Investigative Center, Sinaloa
- Netherlands (5):
  - AURORA Investigative Center, Amsterdam
  - AURORA Investigative Center, Groningen
  - AURORA Investigative Center, Leiden
  - AURORA Investigative Center, Maastricht
  - AURORA Investigative Center, Rotterdam
- AURORA Investigative Center, Skopje, North Macedonia
- Peru (2):
  - AURORA Investigative Center, Lima
  - AURORA Investigative Center, Trujillo
- Philippines (5):
  - AURORA Investigative Center, Angeles City
  - AURORA Investigative Center, Davao City
  - AURORA Investigative Center, Lipa
  - AURORA Investigative Center, Manila
  - AURORA Investigative Center, Quezon City
- Poland (3):
  - AURORA Investigative Center, Katowice
  - AURORA Investigative Center, Warsaw
  - AURORA Investigative Center, Wroclaw
- AURORA Investigative Center, San Juan, Puerto Rico
- Russia (13):
  - AURORA Investigative Center, Kazan'
  - AURORA Investigative Center, Kemerovo
  - AURORA Investigative Center, Krasnoyarsk
  - AURORA Investigative Center, Moscow
  - AURORA Investigative Center, Omsk
  - AURORA Investigative Center, Petrozavodsk
  - AURORA Investigative Center, Rostov-on-Don
  - AURORA Investigative Center, Saint Petersburg
  - AURORA Investigative Center, Samara
  - AURORA Investigative Center, Saratov
  - AURORA Investigative Center, Tolyatti
  - AURORA Investigative Center, Yaroslavl
  - AURORA Investigative Center, Yekaterinburg
- Serbia (2):
  - AURORA Investigative Center, Belgrade
  - AURORA Investigative Center, Niš
- South Africa (4):
  - AURORA Investigative Center, Cape Town
  - AURORA Investigative Center, Johannesburg
  - AURORA Investigative Center, Pretoria
  - AURORA Investigative Center, Stellenbosch
- South Korea (4):
  - AURORA Investigative Center, Daejeon
  - AURORA Investigative Center, Seoul
  - AURORA Investigative Center, Suwon
  - AURORA Investigative Center, Wŏnju
- Spain (4):
  - AURORA Investigative Center, A Coruña
  - AURORA Investigative Center, Barcelona
  - AURORA Investigative Center, Madrid
  - AURORA Investigative Center, Valencia
- Taiwan (3):
  - AURORA Investigative Center, Chang-hua
  - AURORA Investigative Center, Taichung
  - AURORA Investigative Center, Taoyuan District
- Thailand (3):
  - AURORA Investigative Center, Bangkok
  - AURORA Investigative Center, Chiang Mai
  - AURORA Investigative Center, Songkhla
- Turkey (Türkiye) (8):
  - AURORA Investigative Center, Balcalı
  - AURORA Investigative Center, Bursa
  - AURORA Investigative Center, Efeler
  - AURORA Investigative Center, Fatih
  - AURORA Investigative Center, Istanbul
  - AURORA Investigative Center, Konyaalti
  - AURORA Investigative Center, Malatya
  - AURORA Investigative Center, Yenimahalle
- Ukraine (6):
  - AURORA Investigative Center, Kharkiv
  - AURORA Investigative Center, Kyiv
  - AURORA Investigative Center, Lutsk
  - AURORA Investigative Center, Odesa
  - AURORA Investigative Center, Vinnytsia
  - AURORA Investigative Center, Zaporizhzhya
- Vietnam (2):
  - AURORA Investigative Center, Hanoi
  - AURORA Investigative Center, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rovin BH, Parikh SV, Hebert LA, Chan TM, Mok CC, Ginzler EM, Hooi LS, Brunetta P, Maciuca R, Solomons N. Lupus nephritis: induction therapy in severe lupus nephritis--should MMF be considered the drug of choice? Clin J Am Soc Nephrol. 2013 Jan;8(1):147-53. doi: 10.2215/CJN.03290412. Epub 2012 Aug 9. PMID 22879439
- [Background] Ling SY, Huizinga RB, Mayo PR, Larouche R, Freitag DG, Aspeslet LJ, Foster RT. Cytochrome P450 3A and P-glycoprotein drug-drug interactions with voclosporin. Br J Clin Pharmacol. 2014 Jun;77(6):1039-50. doi: 10.1111/bcp.12309. PMID 24330024
- [Background] Ling SY, Huizinga RB, Mayo PR, Freitag DG, Aspeslet LJ, Foster RT. Pharmacokinetics of voclosporin in renal impairment and hepatic impairment. J Clin Pharmacol. 2013 Dec;53(12):1303-12. doi: 10.1002/jcph.166. Epub 2013 Oct 8. PMID 23996158
- [Background] Mayo PR, Huizinga RB, Ling SY, Freitag DG, Aspeslet LJ, Foster RT. Voclosporin food effect and single oral ascending dose pharmacokinetic and pharmacodynamic studies in healthy human subjects. J Clin Pharmacol. 2013 Aug;53(8):819-26. doi: 10.1002/jcph.114. Epub 2013 Jun 4. PMID 23736966
- [Result] Dooley MA, Jayne D, Ginzler EM, Isenberg D, Olsen NJ, Wofsy D, Eitner F, Appel GB, Contreras G, Lisk L, Solomons N; ALMS Group. Mycophenolate versus azathioprine as maintenance therapy for lupus nephritis. N Engl J Med. 2011 Nov 17;365(20):1886-95. doi: 10.1056/NEJMoa1014460. PMID 22087680
- [Result] Busque S, Cantarovich M, Mulgaonkar S, Gaston R, Gaber AO, Mayo PR, Ling S, Huizinga RB, Meier-Kriesche HU; PROMISE Investigators. The PROMISE study: a phase 2b multicenter study of voclosporin (ISA247) versus tacrolimus in de novo kidney transplantation. Am J Transplant. 2011 Dec;11(12):2675-84. doi: 10.1111/j.1600-6143.2011.03763.x. Epub 2011 Sep 22. PMID 21943027
- [Derived] Palmer BF, Tumlin JA, Radhakrishnan J, Rehaume LM, Cross JL, Huizinga RB. The kidney injury biomarker profile of patients with lupus nephritis remains unchanged with the second-generation calcineurin inhibitor voclosporin. Front Nephrol. 2025 Mar 17;5:1540471. doi: 10.3389/fneph.2025.1540471. eCollection 2025. PMID 40166657
- [Derived] Menn-Josephy H, Hodge LS, Birardi V, Leher H. Efficacy of Voclosporin in Proliferative Lupus Nephritis with High Levels of Proteinuria. Clin J Am Soc Nephrol. 2024 Mar 1;19(3):309-318. doi: 10.2215/CJN.0000000000000297. Epub 2023 Dec 18. PMID 38110196
- [Derived] Rovin BH, Teng YKO, Ginzler EM, Arriens C, Caster DJ, Romero-Diaz J, Gibson K, Kaplan J, Lisk L, Navarra S, Parikh SV, Randhawa S, Solomons N, Huizinga RB. Efficacy and safety of voclosporin versus placebo for lupus nephritis (AURORA 1): a double-blind, randomised, multicentre, placebo-controlled, phase 3 trial. Lancet. 2021 May 29;397(10289):2070-2080. doi: 10.1016/S0140-6736(21)00578-X. Epub 2021 May 7. PMID 33971155

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible subjects were randomized in a ratio of 1:1 to receive either voclosporin 23.7 mg twice daily (BID) or matching placebo for 52 weeks. All subjects were also to receive 2 g/day mycophenolate mofetil (MMF). In addition, all subjects were to receive 0.5 g/day intravenous (IV) methylprednisolone on Days 1 and 2 before changing to a reducing course of oral corticosteroid therapy on Day 3.
Groups:
- Voclosporin: Voclosporin 23.7 mg BID + Mycophenolate Mofetil + corticosteroid
- Placebo: Placebo 23.7 mg BID + Mycophenolate Mofetil + corticosteroid
Period: Overall Study
Arm/Group | Voclosporin | Placebo
Started | 179 | 178
Week 24 | 167 | 162
Week 52 | 162 | 147
Completed | 163 | 147
Not Completed | 16 | 31
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 5
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 1 | 3
Not completed — Physician Decision | 2 | 3
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 7 | 14
Not completed — Prohibited medication required | 1 | 0
Not completed — Protocol non-compliance | 1 | 1
Not completed — None of the above | 0 | 4
Not completed — Adverse Event (AE) Prior to First Dose | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat is comprised of all subjects who were randomized treatment, and was used for analysis of all Outcome Measures. Safety population comprised all randomized subjects who took at least one dose of study treatment, and was used for AE and SAE reporting. 1 Voclosporin subject was withdrawn due to an adverse event (AE) prior to receiving the first dose of Voclosporin.
Groups:
- Voclosporin: oral, 23.7 mg BID
  Voclosporin: calcineurin inhibitor
- Placebo: Voclosporin placebo, oral, 3 capsules BID
  Placebo: matching placebo capsule
- Total: Total of all reporting groups
Arm/Group | Voclosporin | Placebo | Total
Number analyzed (Participants) | 179 | 178 | 357
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (10.93) | 33.6 (11) | 33.2 (10.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 152 | 313
  Male | 18 | 26 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 57 | 59 | 116
  Not Hispanic or Latino | 122 | 118 | 240
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 4 | 4
  Asian | 53 | 56 | 109
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 13 | 34
  White | 68 | 61 | 129
  More than one race | 37 | 44 | 81
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — South Africa is included in the Europe count
  participants
    United States | 26 | 26 | 52
    Southeast Asia | 52 | 52 | 104
    Europe | 52 | 52 | 104
    South America | 49 | 48 | 97
Lupus Nephritis (LN) history [Mean (Standard Deviation); unit: years] — Number of years since diagnosis of systemic lupus erythematosus (SLE), lupus nephritis (LN) and first significant proteinuria
  years
    Years since diagnosis of systemic lupus erythematosus (SLE) | 6.6 (6.41) | 6.9 (6.07) | 6.7 (6.23)
    Years since diagnosis of LN | 4.6 (5.07) | 4.7 (4.89) | 4.6 (4.97)
    Years since first Proteinuria | 4.8 (5.2) | 4.6 (4.51) | 4.7 (4.86)
Baseline Urine Protein Creatinine Ratio (UPCR) [Median (Standard Deviation); unit: mg/mg] — Baseline Urine Protein Creatinine Ratio (UPCR) (Average of pre-randomisation values)
  mg/mg | 4.14 (2.711) | 3.87 (2.363) | 4.00 (2.537)
Baseline estimated glomerular filtration rate (eGFR) [Median (Standard Deviation); unit: mL/min/1.73 m2] — Baseline estimated Glomerular Filtration Rate Chronic Kidney Disease Epidemiology Collaboration (CKD-Epi formula) (lowest pre-randomisation value)
  mL/min/1.73 m2 | 92.1 (30.06) | 90.4 (28.97) | 91.2 (29.51)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adjudicated Renal Response at Week 52
Description: The primary efficacy endpoint was the number of subjects showing renal response at Week 52. Renal response was adjudicated based on blinded data by an independent Clinical Endpoints Committee based on meeting the following criteria
  * UPCR of ≤0.5 mg/mg &
  * eGFR ≥60 mL/min/1.73 m2 or no confirmed decrease from baseline in eGFR of >20% &
  * Received no rescue medication for LN &
  * Did not receive more than 10 mg prednisone for ≥3 consecutive days or for ≥7 days in total during Weeks 44 through 52, prior to assessment Note:To be disqualified from renal response, the subject had to fail both eGFR measures (i.e., confirmed eGFR <60 mL/min/1.73 m2 & confirmed >20% drop from baseline) & have an associated treatment-related or disease-related AE that impacted eGFR Withdrawals prior to Week 52 with insufficient Week 52 data to determine response were defined non responders. Subjects who discontinued study drug but continued to attend study visits had their data assessed for response
Time Frame: 52 Weeks
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Oral Capsule: Voclosporin placebo, oral, 3 capsules BID
  Placebo Oral Capsule: matching placebo capsule
Arm/Group | Voclosporin | Placebo Oral Capsule
Number analyzed (Participants) | 179 | 178
Participants
  Number of renal responders | 73 | 40
  Number of renal non-responders | 106 | 138
Statistical Analysis 1: Comparison: Voclosporin vs Placebo Oral Capsule; The primary endpoint was the proportion of subjects showing renal response at Week 52 as adjudicated by the Clinical Endpoints Committee; Test type: Superiority; p < 0.001, Regression, Logistic; The model is based on a logistic regression with terms for treatment, baseline UPCR, biopsy class, MMF use at baseline and Region; Odds Ratio (OR) = 2.65, 95% CI 2-sided [1.64 to 4.27]

2. Secondary Outcome: Number of Participants With Reduction in Urine Protein Creatinine Ratio to 0.5 mg/mg or Less
Description: Number of Participants With Reduction in Urine Protein Creatinine Ratio to 0.5 mg/mg or Less
Time Frame: 52 Weeks
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Oral Capsule: Placebo 23.7 mg BID + Mycophenolate Mofetil + corticosteroid
Arm/Group | Voclosporin | Placebo Oral Capsule
Number analyzed (Participants) | 179 | 178
Participants
  Subjects with UPCR ≤ 0.5 | 116 | 78
  Subjects without UPCR ≤ 0.5 | 63 | 100
Statistical Analysis 1: Comparison: Voclosporin vs Placebo Oral Capsule; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 2.02, 95% CI 2-sided [1.51 to 2.7]

3. Secondary Outcome: Time to Urine Protein Creatinine Ratio of ≤0.5 mg/mg (Number of Days)
Description: Time in days to reduction in Urine Protein Creatinine Ratio to decrease to 0.5 mg/mg or less.
Time Frame: 52 Weeks
Population: Intent to Treat
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Voclosporin | Placebo Oral Capsule
Number analyzed (Participants) | 179 | 178
days | 169 [141 to 214] | 372 [295 to NA] — Upper limit not calculated due to censored data

4. Secondary Outcome: Number of Participants With Renal Response at Week 24
Description: Number of subjects showing renal response at Week 24. Renal response was adjudicated based on blinded data by an Independent Clinical Endpoints Committee based on the following criteria:
  UPCR of ≤0.5 mg/mg, & eGFR ≥60 mL/min/1.73 m2 or no confirmed decrease from baseline in eGFR of >20%, and Received no rescue medication for LN & Did not receive more than 10 mg prednisone for ≥3 consecutive days or for ≥7 days in total during Weeks 16 through 24, just prior to the renal response assessment. Note:To be disqualified from renal response, the subject had to fail both eGFR measures (i.e., confirmed eGFR <60 mL/min/1.73 m2 AND confirmed >20% drop from BL) & have an associated treatment-related or disease-related AE that impacted eGFR. Subjects who withdrew prior to the Week 24 assessment and provided insufficient Week 24 data to determine response were defined as non-responders. Subjects who discontinued study drug but continued to attend study visits had their data assessed for response.
Time Frame: Week 24
Population: intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Voclosporin | Placebo Oral Capsule
Number analyzed (Participants) | 179 | 178
Participants
  Number of renal responders | 58 | 35
  Number of renal non-responders | 121 | 143
Statistical Analysis 1: Comparison: Voclosporin vs Placebo Oral Capsule; Test type: Superiority; p = 0.002, Regression, Cox; Odds Ratio (OR) = 2.23, 95% CI 2-sided [1.34 to 3.72] — The hazard ratios are from a Cox's proportional hazards model with terms for treatment arm, baseline UPCR, biopsy class, MMF use at baseline and Region

5. Secondary Outcome: Number of Subjects With Partial Renal Response at Weeks 24 & 52
Description: Number of subjects with partial Renal Response (defined as a 50% reduction in UPCR from baseline) at Week 24 and at Week 52. Baseline UPCR is the average of 2 pre-randomisation values.
Time Frame: Weeks 24 and 52
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Voclosporin | Placebo Oral Capsule
Number analyzed (Participants) | 179 | 178
Participants
  Week 24 | 126 | 89
  Week 52 | 125 | 92
Statistical Analysis 1: Comparison: Voclosporin vs Placebo Oral Capsule; Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — Week 24; Odds Ratio (OR) = 2.43, 95% CI 2-sided [1.56 to 3.79] — Week 24
Statistical Analysis 2: Comparison: Voclosporin vs Placebo Oral Capsule; Week 52; Test type: Superiority; p < 0.001, Regression, Logistic — Week 52; Odds Ratio (OR) = 2.26, 95% CI 2-sided [1.45 to 3.51] — Week 52

6. Secondary Outcome: Number of Subjects Achieving, and Remaining in, Renal Response (Urine Protein Creatinine Ratio ≤0.5 mg/mg)
Description: Number of subjects achieving, and remaining in, renal response (Urine Protein Creatinine ratio ≤0.5 mg/mg)
Time Frame: Week 52
Population: Intent to Treat population achieving UPCR <0.5 mg/mg
Measure: Count of Participants; unit: Participants
Arm/Group | Voclosporin | Placebo Oral Capsule
Number analyzed (Participants) | 179 | 178
Participants
  Subjects achieving UPCR ≤ 0.5 mg/mg | 116 | 78
  number with 2nd occurrence of UPCR > 0.5 mg/mg | 53 | 37
  number without 2nd occurrence of UPCR > 0.5 mg/mg | 63 | 41
Statistical Analysis 1: Comparison: Voclosporin vs Placebo Oral Capsule; Test type: Superiority; p = 0.349, Regression, Cox; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.53 to 1.25]
Statistical Analysis 2: Comparison: Voclosporin vs Placebo Oral Capsule; Test type: Superiority; p = 0.646, Log Rank

7. Secondary Outcome: Duration of Renal Response (Number of Days)
Description: Duration in days until second occurrence of UPCR >0.5 mg/mg in those subjects who achieve a reduction in UPCR to below 0.5 mg/mg
Time Frame: Week 52
Population: Intent to Treat
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Voclosporin | Placebo Oral Capsule
Number analyzed (Participants) | 116 | 78
days | 216 [127 to NA] — Upper limit not calculated due to censored data | 198 [103 to NA] — Upper limit not calculated due to censored data

8. Secondary Outcome: Number of Subjects Achieving 50% Reduction in Urine Protein Creatinine Ratio
Description: Number of subjects achieving 50% reduction in Urine Protein Creatinine ratio
Time Frame: 52 Weeks
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Voclosporin | Placebo Oral Capsule
Number analyzed (Participants) | 179 | 178
Participants
  Subjects with 50% UPCR reduction | 173 | 135
  Subjects without 50% UPCR reduction | 6 | 43

9. Secondary Outcome: Time to 50% Reduction in UPCR (Number of Days)
Description: Time in days to reduction in Urine Protein Creatinine Ratio to decrease by 50% compared to baseline. Baseline is the average of two pre-randomisation values.
Time Frame: 52 weeks
Population: Intent to Treat
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Voclosporin | Placebo Oral Capsule
Number analyzed (Participants) | 179 | 178
days | 29 [29 to 32] | 63 [57 to 87]
Statistical Analysis 1: Comparison: Voclosporin vs Placebo Oral Capsule; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 2.05, 95% CI 2-sided [1.62 to 2.6]

10. Secondary Outcome: Change From Baseline in eGFR
Description: Change from baseline by visit in estimated Glomerular Filtration rate. eGFR is corrected to a maximum value of 90 mL/min/1.73 m2
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 16, 20, 24, 30, 36, 42, 48 and 52.
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: ml/min/1.73 square metres
Arm/Group | Voclosporin | Placebo Oral Capsule
Number analyzed (Participants) | 179 | 178
ml/min/1.73 square metres
  Baseline | 78.3 (15.83) | 77.4 (16.98)
  Week 2 change from baseline | -1.5 (9.44) | 3.3 (10.12)
  Week 4 change from baseline | -0.4 (10.39) | 3.2 (9.86)
  Week 8 change from baseline | -0.9 (13.1) | 3.8 (11.27)
  Week 12 change from baseline | -0.3 (11.74) | 3.3 (12.85)
  Week 16 change from baseline | -0.1 (12.27) | 2.8 (13.25)
  Week 20 change from baseline | -0.7 (12.09) | 3.2 (13.04)
  Week 24 change from baseline | -0.3 (13.8) | 2.8 (13.84)
  Week 30 change from baseline | -0.8 (14.2) | 1.8 (14.4)
  Week 36 change from baseline | -1.9 (14.89) | 1.5 (14.84)
  Week 42 change from baseline | -2.8 (16.7) | 1.5 (15.53)
  Week 48 change from baseline | -3.6 (17.2) | 1.1 (15.71)
  Week 52 change from baseline | -1.5 (16.16) | 1.5 (15)
Statistical Analysis 1: Comparison: Voclosporin vs Placebo Oral Capsule; Week 2; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Least Squares) = -4.6, 95% CI 2-sided [-7.3 to -1.9], Standard Error of Mean 1.39
Statistical Analysis 2: Comparison: Voclosporin vs Placebo Oral Capsule; Week 4; Test type: Superiority; p = 0.014, Mixed Models Analysis; Mean Difference (Least Squares) = -3.4, 95% CI 2-sided [-6.1 to -0.7], Standard Error of Mean 1.39
Statistical Analysis 3: Comparison: Voclosporin vs Placebo Oral Capsule; Week 8; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Least Squares) = -4.6, 95% CI 2-sided [-7.3 to -1.9], Standard Error of Mean 1.39
Statistical Analysis 4: Comparison: Voclosporin vs Placebo Oral Capsule; Week 12; Test type: Superiority; p = 0.017, Mixed Models Analysis; Mean Difference (Least Squares) = -3.3, 95% CI 2-sided [-6 to -0.6], Standard Error of Mean 1.39
Statistical Analysis 5: Comparison: Voclosporin vs Placebo Oral Capsule; Week 16; Test type: Superiority; p = 0.085, Mixed Models Analysis; Mean Difference (Least Squares) = -2.4, 95% CI 2-sided [-5.1 to 0.3], Standard Error of Mean 1.4
Statistical Analysis 6: Comparison: Voclosporin vs Placebo Oral Capsule; Week 20; Test type: Superiority; p = 0.035, Mixed Models Analysis; Mean Difference (Least Squares) = -3, 95% CI 2-sided [-5.7 to -0.2], Standard Error of Mean 1.4
Statistical Analysis 7: Comparison: Voclosporin vs Placebo Oral Capsule; Week 24; Test type: Superiority; p = 0.121, Mixed Models Analysis; Mean Difference (Least Squares) = -2.2, 95% CI 2-sided [-5 to 0.6], Standard Error of Mean 1.41
Statistical Analysis 8: Comparison: Voclosporin vs Placebo Oral Capsule; Week 30; Test type: Superiority; p = 0.12, Mixed Models Analysis; Mean Difference (Least Squares) = -2.2, 95% CI 2-sided [-5 to 0.6], Standard Error of Mean 1.42
Statistical Analysis 9: Comparison: Voclosporin vs Placebo Oral Capsule; Week 36; Test type: Superiority; p = 0.102, Mixed Models Analysis; Mean Difference (Least Squares) = -2.3, 95% CI 2-sided [-5.1 to 0.5], Standard Error of Mean 1.43
Statistical Analysis 10: Comparison: Voclosporin vs Placebo Oral Capsule; Week 42; Test type: Superiority; p = 0.022, Mixed Models Analysis; Mean Difference (Least Squares) = -3.3, 95% CI 2-sided [-6.1 to 0.5], Standard Error of Mean 1.44
Statistical Analysis 11: Comparison: Voclosporin vs Placebo Oral Capsule; Week 48; Test type: Superiority; p = 0.004, Mixed Models Analysis; Mean Difference (Least Squares) = -4.1, 95% CI 2-sided [-7 to -1.3], Standard Error of Mean 1.45
Statistical Analysis 12: Comparison: Voclosporin vs Placebo Oral Capsule; Week 52; Test type: Superiority; p = 0.055, Mixed Models Analysis; Mean Difference (Least Squares) = -2.8, 95% CI 2-sided [-5.7 to 0.1], Standard Error of Mean 1.46

11. Secondary Outcome: Change From Baseline in UPCR
Description: Change from baseline by visit in Urine Protein Creatinine Ratio. Baseline is the average of two pre-randomisation values.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 16, 20, 24, 30, 36, 42, 48 and 52.
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mg/mg
Arm/Group | Voclosporin | Placebo Oral Capsule
Number analyzed (Participants) | 179 | 178
mg/mg
  Baseline | 4.14 (2.711) | 3.87 (2.363)
  Week 2 change from baseline | -1.46 (1.991) | -0.7 (2.312)
  Week 4 change from baseline | -1.98 (2.29) | -1.07 (2.155)
  Week 8 change from baseline | -2.23 (2.213) | -1.43 (2.448)
  Week 12 change from baseline | -2.56 (2.293) | -1.48 (2.688)
  Week 16 change from baseline | -2.75 (2.462) | -1.58 (2.81)
  Week 20 change from baseline | -2.74 (2.968) | -1.54 (2.82)
  Week 24 change from baseline | -2.74 (2.567) | -1.59 (2.899)
  Week 30 change from baseline | -2.66 (3.336) | -1.7 (3.112)
  Week 36 change from baseline | -2.74 (2.871) | -1.63 (3.188)
  Week 42 change from baseline | -2.91 (2.522) | -1.78 (3.39)
  Week 48 change from baseline | -2.71 (2.807) | -1.8 (3.004)
  Week 52 change from baseline | -2.65 (2.872) | -1.88 (3.05)
Statistical Analysis 1: Comparison: Voclosporin vs Placebo Oral Capsule; Week 2; Test type: Superiority; p = 0.011, Mixed Models Analysis; Mean Difference (Least Squares) = -0.56, 95% CI 2-sided [-1 to -0.13], Standard Error of Mean 0.181
Statistical Analysis 2: Comparison: Voclosporin vs Placebo Oral Capsule; Week 4; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Least Squares) = -0.76, 95% CI 2-sided [-1.13 to -0.4], Standard Error of Mean 0.187
Statistical Analysis 3: Comparison: Voclosporin vs Placebo Oral Capsule; Week 8; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Least Squares) = -0.7, 95% CI 2-sided [-1.05 to -0.34], Standard Error of Mean 0.181
Statistical Analysis 4: Comparison: Voclosporin vs Placebo Oral Capsule; Week 12; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Least Squares) = -0.94, 95% CI 2-sided [-1.33 to -0.55], Standard Error of Mean 0.196
Statistical Analysis 5: Comparison: Voclosporin vs Placebo Oral Capsule; Week 16; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Least Squares) = -1.18, 95% CI 2-sided [-1.6 to -0.76], Standard Error of Mean 0.214
Statistical Analysis 6: Comparison: Voclosporin vs Placebo Oral Capsule; Week 20; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Least Squares) = -1.16, 95% CI 2-sided [-1.63 to -0.68], Standard Error of Mean 0.241
Statistical Analysis 7: Comparison: Voclosporin vs Placebo Oral Capsule; Week 24; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Least Squares) = -1.15, 95% CI 2-sided [-1.59 to -0.72], Standard Error of Mean 0.222
Statistical Analysis 8: Comparison: Voclosporin vs Placebo Oral Capsule; Week 30; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Least Squares) = -1.02, 95% CI 2-sided [-1.58 to -0.46], Standard Error of Mean 0.284
Statistical Analysis 9: Comparison: Voclosporin vs Placebo Oral Capsule; Week 36; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Least Squares) = -1.21, 95% CI 2-sided [-1.73 to -0.69], Standard Error of Mean 0.264
Statistical Analysis 10: Comparison: Voclosporin vs Placebo Oral Capsule; Week 42; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Least Squares) = -1.37, 95% CI 2-sided [-1.87 to -0.86], Standard Error of Mean 0.256
Statistical Analysis 11: Comparison: Voclosporin vs Placebo Oral Capsule; Week 48; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Least Squares) = -1.06, 95% CI 2-sided [-1.56 to -0.55], Standard Error of Mean 0.256
Statistical Analysis 12: Comparison: Voclosporin vs Placebo Oral Capsule; Week 52; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Least Squares) = -0.99, 95% CI 2-sided [-1.52 to -0.46], Standard Error of Mean 0.27

12. Secondary Outcome: Number of Subjects With Renal Response With Low Dose Steroids
Description: Programmed Renal Response whilst on low dose steroids (<2.5 mg/day) for the preceding 8 Weeks at Weeks 24 and 52
Time Frame: Week 24 and Week 52
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Voclosporin | Placebo Oral Capsule
Number analyzed (Participants) | 179 | 178
Participants
  Renal Response at Week 24 | 32 | 16
  Renal Response at Week 52 | 64 | 36
Statistical Analysis 1: Comparison: Voclosporin vs Placebo Oral Capsule; Week 24; Test type: Superiority; p = 0.008, Regression, Logistic — Week 24; Odds Ratio (OR) = 2.44, 95% CI 2-sided [1.26 to 4.71] — Week 24
Statistical Analysis 2: Comparison: Voclosporin vs Placebo Oral Capsule; Week 52; Test type: Superiority; p < 0.001, Regression, Logistic — Week 52; Odds Ratio (OR) = 2.44, 95% CI 2-sided [1.48 to 4.00] — Week 52

13. Secondary Outcome: Change From Baseline in Safety of Estrogens in Systemic Lupus Erythematosus National Assessment Systemic Lupus Erythematosus Disease Activity Index (SELENA - SLEDAI)
Description: Change from baseline in Safety of Estrogens in Systemic Lupus Erythematosus National Assessment Systemic Lupus Erythematosus Disease Activity Index (SELENA-SLEDAI) score at Week 24 and 52.
  The SELENA-SLEDAI tool is a cumulative and weighted index used to assess disease activity across 24 different disease descriptors in patients with lupus. A patient's SELENA-SLEDAI total score is the sum of all marked lupus related descriptors (seizure, psychosis, organic brain syndrome, visual disturbance, cranial nerve disorder, lupus headache, cerebrovascular accident, vasculitis, arthritis, myositis, urinary casts, hematuria, proteinuria, pyuria, new rash, alopecia, mucosal ulcers, pleurisy, pericarditis, low complement, increased DNA binding, fever, thrombocytopenia, leukopenia). A total score can fall between 0 and 105, with a higher score representing a more significant degree of disease activity.
Time Frame: Week 24 and Week 52
Population: Intent to Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Voclosporin | Placebo Oral Capsule
Number analyzed (Participants) | 179 | 178
scores on a scale
  Change from baseline at Week 24 | -4.5 [-5.4 to -3.7] | -4.1 [-5.0 to -3.2]
  Change from baseline at Week 52 | -6 [-6.7 to -5.2] | -5.5 [-6.3 to -4.7]
Statistical Analysis 1: Comparison: Voclosporin vs Placebo Oral Capsule; Week 24; Test type: Superiority; p = 0.373, Mixed Models Analysis — Week 24; Least Squares Mean difference = -0.5, 95% CI 2-sided [-1.6 to 0.6] — Week 24
Statistical Analysis 2: Comparison: Voclosporin vs Placebo Oral Capsule; Week 52; Test type: Superiority; p = 0.277, Mixed Models Analysis — Week 52; Least Squares Mean difference = -0.5, 95% CI 2-sided [-1.4 to 0.4] — Week 52

14. Secondary Outcome: Change From Baseline in Patient Reported Outcomes
Description: Health-related quality of life (HRQoL) information was collected using the Short Form Health Survey (SF-36) HRQoL assessment and the LupusPRO (v1.7) assessment.
  The SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. Scoring ranges from 0 to 100 with higher scores reflecting better health.
  LupusPro assessment is a patient-reported questionnaire regarding the effect of lupus or its treatment on the patient's health, quality of life, and the medical care received related to lupus. The questionnaire consists of 43 questions within 8 HRQOL domains and 4 Non-HRQoL domains. Scores range from 0 to 100 with higher scores reflecting better quality of life.
Time Frame: Week 24 and Week 52
Population: Intent to Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Voclosporin | Placebo Oral Capsule
Number analyzed (Participants) | 179 | 178
score on a scale
  SF-36 change from baseline at Week 24 | 6.64 [4.34 to 8.93] | 7.11 [4.80 to 9.42]
  SF-36 change from baseline at Week 52 | 10.44 [8.04 to 12.83] | 10.81 [8.37 to 13.25]
  LupusPRO HRQOL change from baseline at Week 24 | 7.7 [5.40 to 10.13] | 6.06 [3.68 to 8.45]
  LupusPRO HRQOL change from baseline at Week 52 | 9.24 [6.78 to 11.70] | 9.84 [7.33 to 12.35]
  LupusPRO non-HRQOL change from baseline at Week 24 | 1.06 [-1.32 to 3.44] | 2.94 [0.54 to 5.35]
  LupusPRO non-HRQOL change from baseline at Week 52 | 4.08 [1.60 to 6.56] | 3.74 [1.22 to 6.26]
Statistical Analysis 1: Comparison: Voclosporin vs Placebo Oral Capsule; SF-36 Change from Baseline Week 24; Test type: Superiority; p = 0.733, Mixed Models Analysis; Slope = -0.47, 95% CI 2-sided [-3.21 to 2.26], Standard Error of Mean 1.389
Statistical Analysis 2: Comparison: Voclosporin vs Placebo Oral Capsule; SF-36 Change from Baseline at Week 52; Test type: Superiority; p = 0.801, Mixed Models Analysis; Mean Difference (Least Squares) = -0.37, 95% CI 2-sided [-3.29 to 2.54], Standard Error of Mean 1.481
Statistical Analysis 3: Comparison: Voclosporin vs Placebo Oral Capsule; LupusPRO HRQOL Change from Baseline at Week 24; Test type: Superiority; p = 0.239, Mixed Models Analysis; Mean Difference (Least Squares) = 1.7, 95% CI 2-sided [-1.14 to 4.54], Standard Error of Mean 1.442
Statistical Analysis 4: Comparison: Voclosporin vs Placebo Oral Capsule; LupusPRO HRQOL Change from Baseline at Week 52; Test type: Superiority; p = 0.695, Mixed Models Analysis; Mean Difference (Least Squares) = -0.6, 95% CI 2-sided [-3.62 to 2.42], Standard Error of Mean 1.535
Statistical Analysis 5: Comparison: Voclosporin vs Placebo Oral Capsule; LupusPRO non-HRQOL Change from Baseline at Week 24; Test type: Superiority; p = 0.19, Mixed Models Analysis; Mean Difference (Least Squares) = -1.89, 95% CI 2-sided [-4.72 to 0.94], Standard Error of Mean 1.439
Statistical Analysis 6: Comparison: Voclosporin vs Placebo Oral Capsule; LupusPRO non-HRQOL Change from Baseline at Week 52; Test type: Superiority; p = 0.826, Mixed Models Analysis; Mean Difference (Least Squares) = 0.826, 95% CI 2-sided [-2.67 to 3.35], Standard Error of Mean 1.531

ADVERSE EVENTS:
Time Frame: Reporting period is from first dose up to 30 days following last dose (Week 52).
Description: Treatment emergent Deaths and serious adverse events (SAEs). Reporting period is from first dose up to 30 days following last dose
Arm/Group | Voclosporin | Placebo Oral Capsule
All-Cause Mortality (participants affected / at risk) | 1/178 | 5/178
Serious Adverse Events (participants affected / at risk) | 37/178 | 38/178
Other Adverse Events (participants affected / at risk) | 161/178 | 156/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Voclosporin (N=178) | Placebo Oral Capsule (N=178)
Pneumonia (Infections and infestations) | 7 (8) | 8 (9)
Gastroenteritis (Infections and infestations) | 3 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial diarrhoea (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia cytomegaloviral (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 3 (3)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster disseminated (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Paraspinal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Salmonellosis (Infections and infestations) | 0 (0) | 1 (1)
Salpingitis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 4 (5) | 2 (2)
Renal impairment (Renal and urinary disorders) | 2 (2) | 1 (1)
Lupus nephritis (Renal and urinary disorders) | 1 (1) | 4 (4)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Lupus encephalitis (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Neuropsychiatric lupus (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 2 (3)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lupus pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 1 (1)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Voclosporin (N=178) | Placebo Oral Capsule (N=178)
Upper respiratory tract infection (Infections and infestations) | 31 (44) | 26 (33)
Viral upper respiratory tract infection (Infections and infestations) | 20 (24) | 18 (20)
Urinary tract infection (Infections and infestations) | 17 (25) | 13 (14)
Herpes zoster (Infections and infestations) | 13 (13) | 9 (9)
Influenza (Infections and infestations) | 12 (15) | 10 (12)
Gastroenteritis (Infections and infestations) | 7 (8) | 10 (10)
Pharyngitis (Infections and infestations) | 3 (3) | 9 (11)
Diarrhoea (Gastrointestinal disorders) | 34 (43) | 21 (23)
Abdominal pain upper (Gastrointestinal disorders) | 13 (13) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 10 (11) | 2 (3)
Nausea (Gastrointestinal disorders) | 10 (10) | 17 (18)
Dyspepsia (Gastrointestinal disorders) | 10 (10) | 3 (3)
Vomiting (Gastrointestinal disorders) | 5 (6) | 12 (17)
Glomerular filtration rate decreased (Investigations) | 43 (61) | 15 (19)
Headache (Nervous system disorders) | 29 (34) | 11 (16)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (10) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 17 (20)
Hypertension (Vascular disorders) | 35 (38) | 14 (15)
Oedema peripheral (General disorders) | 11 (11) | 11 (11)
Anaemia (Blood and lymphatic system disorders) | 18 (19) | 10 (11)
Leukopenia (Blood and lymphatic system disorders) | 7 (8) | 10 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 3 (3)
Renal impairment (Renal and urinary disorders) | 11 (14) | 5 (6)
Lupus nephritis (Renal and urinary disorders) | 1 (1) | 8 (8)
Proteinuria (Renal and urinary disorders) | 0 (0) | 8 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol: Protocol V1.0 01Dec2016 (2016-12-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT03021499/Prot_001.pdf
  • Study Protocol: Protocol V2.0 04May2017 (2017-05-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT03021499/Prot_002.pdf
  • Statistical Analysis Plan (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT03021499/SAP_000.pdf